CLINICAL TRIAL: NCT00581919
Title: Phase II Trial of Bortezomib, Low Dose Dexamethasone, and Doxorubicin With Acetyl-L-Carnitine for Neuroprotection in Patients With Previously Treated Multiple Myeloma
Brief Title: Ph 2 Bortezomib, Dexamethasone, + Doxorubicin With ALCAR for Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO04402; H-2004-0064 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2011-00516 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2016-11

CONDITIONS: Multiple Myeloma
Keywords: previously treated multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Doxorubicin; Acetylcarnitine; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bort, Dex, and Dox with ALCAR (Experimental)
  Interventions: Drug: Bort, Dex, and Dox with ALCAR

INTERVENTIONS:
Drug: Bort, Dex, and Dox with ALCAR — Bortezomib 1.3 mg/m2 IV days 1, 4, 8, and 11 Dexamethasone 20 mg PO days 1, 4, 8, and 11 Doxorubicin 15 mg/m2 IV days 1 and 8 Acetyl-L-Carnitine (ALCAR) 1.5 g PO BID days 1-21 Maximum of 8 cycles. Each cycle is 21 days long
  Other Names: Velcade, cc-5013, ALCAR

SUMMARY:
Patients will receive Bortezomib, Dexamethasone, and Doxorubicin in 21 day cycles a total of 4 to 8 times (based on response to the treatment). Patients will also receive acetyl-L-carnitine (ALCAR) daily.

DETAILED DESCRIPTION:
The primary objective of this study is to assess overall response rate to the treatment.

Secondary objectives include: evaluating and describing the incidence of chemotherapy-induced peripheral neuropathy using the FACT/GOG-Ntx assessment tool; evaluating the utility of adding ALCAR to the chemotherapy to reduce the incidence of peripheral neuropathy; and evaluating the utility of the Grooved Pegboard Completion Time as a longitudinal measure of peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated multiple myeloma with measurable serum or urine monoclonal protein.

Exclusion Criteria:

* Patients with previous doxorubicin treatment totaling 220 mg/m2 or more
* LVEF less than 45%
* Patients with >grade II sensory neuropathy at baseline as assessed by the PI will be excluded
* No history of seizures as ALCAR may lower the seizure threshold
* Known HIV infection
* Current pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-02; Primary Completion 2010-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie S Callander, MD, Principal Investigator — UWCCC
Locations (5):
- United States (5):
  - Mercy Health Systems, Janesville, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Cancer Center, Madison, Wisconsin
  - Regional Cancer Center, Waukesha/Oconomowoc, Wisconsin
  - Aspirus Wausau Hospital, Aspirus Regional Cancer Center, Wausau, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of Wisconsin Hospital and Clinics and the Wisconsin Oncology Network between April 2004 and September 2010.
Pre-assignment Details: No events between enrollment and group assignment. All subjects are enrolled are assigned to the same group.
Period: Overall Study
Arm/Group | Bort, Dex, and Dox With ALCAR
Started | 32
Completed | 8
Not Completed | 24
Not completed — Adverse Event | 8
Not completed — Death | 1
Not completed — Disease Progression | 10
Not completed — Physician Decision | 1
Not completed — Other Complicating Disease | 1
Not completed — Started Non-Protocol Therapy | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bort, Dex, and Dox With ALCAR
Number analyzed (Participants) | 32
Age, Customized [Number; unit: participants]
  30-39 | 1
  40-49 | 4
  50-59 | 6
  60-69 | 12
  70-79 | 7
  80-89 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Anti-tumor Response Rate (Complete Response and Partial Response) to the Combination of Bortezomib, Dexamethasone, Doxorubicin, and ALCAR
Description: Anti-tumor responses were analyzed descriptively and summarized in tabular format. Ninety percent confidence intervals for the percentage of subjects with a confirmed anti-tumor response were constructed using the method proposed by Duffy-Santner.
  Complete response defined as: no evidence of M-protein on immunofixation of serum and/or urine AND less than 5% plasma cells in the bone marrow biopsy.
  Partial response defined as: 50 to 99% decrease in M-protein on serum and/or urine protein electrophoresis.
Time Frame: Every 21 days, up to 24 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bort, Dex, and Dox With ALCAR
Number analyzed (Participants) | 32
percentage of participants | 53 [36 to 69]

2. Secondary Outcome: Overall Survival
Time Frame: From date of randomization until the date of death from any cause, assessed up to 7 years
Measure: Median (Full Range); unit: months
Arm/Group | Bort, Dex, and Dox With ALCAR
Number analyzed (Participants) | 32
months | 28.3 [0.2 to 75.3]

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined as any of the following: 1) 25% or greater increase in M-protein as measured by serum or urine protein electrophoresis. There must be an absolute minimum increase of 0.5 g/dl in serum M spike or 0.2 gram of specific urinary light chains to constitute progression, 2) 25% or greater increase in the percentage or plasma cells in the bone marrow biopsy, or 3) new bone lesions or an increase in the size of old lesions on x-ray.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 years.
Measure: Median (Full Range); unit: months
Arm/Group | Bort, Dex, and Dox With ALCAR
Number analyzed (Participants) | 32
months | 5 [1.0 to 37.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected while subjects were receiving study treatment through 30 days post last dose of study treatment, up to 28 weeks.
Arm/Group | Bort, Dex, and Dox With ALCAR
Serious Adverse Events (participants affected / at risk) | 10/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bort, Dex, and Dox With ALCAR (N=32)
Thrombosis/embolism - DVT (Vascular disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
CNS Hemorrhage/bleeding (Nervous system disorders) | 2
Hemorrhage - Other, specify: GI-esophagus (Gastrointestinal disorders) | 1
Febrile neutropenia - pneumonia (Infections and infestations) | 1
Infection with unknown ANC (Infections and infestations) | 2
Infection without Neutropenia (Infections and infestations) | 1
Infection/Febrile Neutropenia (Infections and infestations) | 1
Infection/Febrile Neutropenia - Other, specify: Normal ANC, Gr 1 or 2 neutrophils (Infections and infestations) | 1
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other, specify: encephalopathy (Nervous system disorders) | 1
Neurology - Other, specify: vocal cord paralysis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bort, Dex, and Dox With ALCAR (N=32)
abdominal pain (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 21
Anorexia (Metabolism and nutrition disorders) | 8
back pain (Musculoskeletal and connective tissue disorders) | 5
Bloating (Gastrointestinal disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Blurred vision (Eye disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 5
Colitis (Gastrointestinal disorders) | 2
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatine increased (Investigations) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 6
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Edema limbs (General disorders) | 9
Extrapyramidal involuntary movement (Nervous system disorders) | 3
Fatigue (General disorders) | 17
Fever (General disorders) | 4
Headache (Nervous system disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Infections and infestations other, specify: with or without neutropenia (Infections and infestations) | 7
Insomnia (Psychiatric disorders) | 7
LDH (Investigations) | 2
Lymphocyte count decrease (Investigations) | 10
Metabolic changes (Metabolism and nutrition disorders) | 2
Muscle pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder- other, specify: Joint pain (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 16
Neuropathic pain (Nervous system disorders) | 7
Neutrophil count decreased (Investigations) | 15
Oral pain (Gastrointestinal disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 22
Platelet count decreased (Investigations) | 23
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Rectal hemorrhage (Gastrointestinal disorders) | 2
Sweating (Skin and subcutaneous tissue disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 5
Upper respiratory infection (Infections and infestations) | 8
Urinary frequency (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 5
White blood cell decreased (Investigations) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No